CLINICAL TRIAL: NCT06306846
Title: Neoadjuvant Stereotactic Body Radiotherapy（SBRT）Combined With Immunotherapy for Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Neoadjuvant SBRT in Localized Advanced HNSCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiang Feng (Other)
Responsible Party: Sponsor-Investigator, Jiang Feng, principal investigator, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11235794
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Head and Neck Squamous Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- experimental (Experimental): Step 1：neoadjuvant anti-PD-1 antibody and TP chemotherapy every 3 weeks 2 cycles
  Step 2： SBRT with GTV expanded 3mm , 24Gy/3F, every other day within one week after the immunochemotherapy
  Step 3：Subsequent surgery and adjuvant treatments.
  Radical surgery will be performed within 4-6 weeks after the second cycle of immunochemotherapy，no matter the situation of the tumor regresses.
  Patients with pathological MPR/CR were treated with PD-1 antibody every two weeks up to 6 cycles after surgery with no adjuvant chemoradiotherapy. Those not achieved MPR/CR will receive adjuvant radiotherapy or chemoradiotherapy according to NCCN guidelines.
  Interventions: Radiation: SBRT+immunochemotherpy
- control (Active Comparator): Step 1：neoadjuvant anti-PD-1 antibody and TP chemotherapy every 3 weeks 2 cycles
  Step 2：Subsequent surgery and adjuvant treatments.
  Radical surgery will be performed within 4-6 weeks after the second cycle of immunochemotherapy，no matter the situation of the tumor regresses.
  Patients with pathological MPR/CR were treated with PD-1 antibody every two weeks up to 6 cycles after surgery without adjuvant chemoradiotherapy. Those not achieved MPR/CR will receive adjuvant radiotherapy or chemoradiotherapy according to NCCN guidelines.
  Interventions: Drug: Immunochemotherapy
- Cetuximab+immunochemo (Active Comparator): Step 1：neoadjuvant anti-PD-1 antibody and TP chemotherapy combined with cetuximab every 3 weeks for 2 cycles
  step2: Subsequent surgery and adjuvant treatments.
  Radical surgery will be performed within 4-6 weeks after the second cycle of immunochemotherapy，no matter the situation of the tumor regresses.
  Patients with pathological MPR/CR were treated with PD-1 antibody and cetuximab every two weeks up to 6 cycles after surgery without adjuvant chemoradiotherapy. Those not achieved MPR/CR will receive adjuvant radiotherapy or chemoradiotherapy according to NCCN guidelines.
  Interventions: Drug: cetuximab+immunochemotharpy

INTERVENTIONS:
Radiation: SBRT+immunochemotherpy — SBRT radiotherapy，followed with PD-1 monoclonal antibody and TP chemotherapy
  Other Names: immunochemotherapy
  Arms: experimental
Drug: Immunochemotherapy — PD-1 monoclonal antibody and TP chemotheapy
  Arms: control
Drug: cetuximab+immunochemotharpy — PD-1 monoclonal antibody and TP chemotheapy combined with cetuximab
  Arms: Cetuximab+immunochemo

SUMMARY:
The response rate of HNSCC to immune checkpoint blockade was not satisfied. Improving the mPR rate of neoadjuvant immunotherapy through the combination with other treatment methods is an important way to further improve the prognosis of such patients. This study aims to explore the efficacy and safety of PD-1 monoclonal antibody with neoadjvant SBRT and chemotherapy. The triple mode not only can Increase the effectiveness of neoadjuvant therapy，meanwhile，the in situ tumor vaccine inoculation effect generated by enhancing the release of specific antigens after tumor radiotherapy with PD-1 monoclonal antibody achieves a sustained anti-tumor immune effect throughout the body， reducing postoperative adjuvant radiotherapy and chemotherapy. The triple mode has important exploratory value in achieving high quality and long-term survival for patients, and may provides a more efficient mode for locally advanced HNSCC.

DETAILED DESCRIPTION:
locally advanced HNSCC patients would receive PD-1 antibody and chemotherapy with or without SBRT covering GTV of primary disease and metastatic nodes , followed by surgery. pathological response was measured .Neoadjuvant PD-1 antibody and chemotherapy with certuxmab was also tested

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed initially resectable Localized advanced head and neck squamous cell carcinoma，and plan for surgical resection.
2. Immunohistochemical confirmed the HPV status through P16 immunostaining.
3. Male or female, Between the aged from 18 to 70 years,
4. Able to provide informed consent, comply with agreements, and sign research specific consent documents.
5. ZPS is less than 2.
6. Adequate bone marrow, liver and kidney, heart , lung and other physiological function determined by Researchers, able to tolerate neoadjuvant anti-PD-1, anti-EGFR, and radiation therapy.
7. Subjects are willing and able to comply with visits, treatment regimens, laboratory tests, and other requirements of the study as spe.

Exclusion Criteria:

1. Any clinical illness, such as hemorrhage, active infection, or mental illness, that can hinder safe participation or adherence of research procedures.
2. Patients who cannot accept radiotherapy in standard treatment.
3. Long term maintenance of oral steroids (≥ 20mg prednisone equivalent per day) is required, excluding patients with inhaled, local, or non absorbable steroids.
4. Autoimmune diseases, including but not limited to inflammatory bowel disease, rheumatoid arthritis, autoimmune hepatitis, systemic sclerosis (scleroderma and variants), systemic lupus erythematosus, autoimmune vasculitis, autoimmune neuropathy (such as Guillain Barre syndrome), etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
major pathology response (MPR) | 4-6 weeks after the end of the neoadjuvant therapy
  major pathology response

CONTACTS AND LOCATIONS:
Overall Officials: feng Jiang, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China